CLINICAL TRIAL: NCT00953511
Title: Prospective Study to Analyze the Predictive Role of Factors Implicated in the Signaling Pathway of ERCC1 in Response to Treatment With Neoadjuvant Radiochemotherapy in Patients With Esophageal Cancer
Brief Title: Cologne Esophageal Response Prediction Study (CERP-Study)
Acronym: CERP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elfriede Bollschweiler (Other)
Responsible Party: Sponsor-Investigator, Elfriede Bollschweiler, Professor of Surgical Research, University of Cologne
Organization: University of Cologne (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UK-09-118
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Esophageal Cancer
Keywords: esophagus; chemoradiation; excision repair cross-complementing gene; polymorphism; response prediction
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- genetic (Other)
  Interventions: Genetic: ERCC1 pathways analysis

INTERVENTIONS:
Genetic: ERCC1 pathways analysis — The gene polymorphism of ERCC1 rs11615 and the pathways of ERRC1 will be analyzed in endoscopic tumor biopsies as well as in normal tissues prior to therapy. The results will be compared with histopathologic response after neoadjuvant therapy.

SUMMARY:
RATIONALE: The prognosis of patients with advanced esophageal cancer may be improved by preoperative chemoradiation. But only those patients have a benefit from this additional therapy, whose tumor shows a response after chemoradiation. Molecular markers may help to identify before starting the therapy those patients who response.

PURPOSE: This is the first prospective, clinical trial to study the impact of ERCC1 to predict histopathological response to neoadjuvant radiochemotherapy (RTx/CTx) in patients with cancer of the esophagus.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* newly diagnosed adenocarcinoma or squamous cell carcinoma of the esophagus or cardia

Exclusion Criteria:

* missing informed consent
* prior radiation or chemotherapy
* second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-08; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
histopathologic response to chemoradiation | 1 month postoperative
  Patients with cT3 esophageal cancer received RTx/CTx according a standardized protocol. 6 weeks after this neoadjuvant therapy a tranthoracic esophagectomy with two-field lymphadenectomy will be performed.
  The histopathologic response is measured using the surgical specimen.

SECONDARY OUTCOMES:
prognosis | 2 years after surgical resection
  All patients get a standardized follow-up every three month evaluating clinical signs of response. If necessary additional diagnostic procedures will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf H. Hölscher, MD, Principal Investigator — Department of General, Visceral and Cancer Surgery, University of Cologne
Locations (1):
- Department of General, Visceral and Cancer Surgery, University of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warnecke-Eberz U, Vallbohmer D, Alakus H, Kutting F, Lurje G, Bollschweiler E, Wienand-Dorweiler A, Drebber U, Holscher AH, Metzger R. ERCC1 and XRCC1 gene polymorphisms predict response to neoadjuvant radiochemotherapy in esophageal cancer. J Gastrointest Surg. 2009 Aug;13(8):1411-21. doi: 10.1007/s11605-009-0881-z. Epub 2009 May 7. PMID 19421825
- [Background] Brabender J, Vallbohmer D, Grimminger P, Hoffmann AC, Ling F, Lurje G, Bollschweiler E, Schneider PM, Holscher AH, Metzger R. ERCC1 RNA expression in peripheral blood predicts minor histopathological response to neoadjuvant radio-chemotherapy in patients with locally advanced cancer of the esophagus. J Gastrointest Surg. 2008 Nov;12(11):1815-21. doi: 10.1007/s11605-008-0668-7. Epub 2008 Sep 3. PMID 18769985
- [Background] Bollschweiler E, Metzger R, Drebber U, Baldus S, Vallbohmer D, Kocher M, Holscher AH. Histological type of esophageal cancer might affect response to neo-adjuvant radiochemotherapy and subsequent prognosis. Ann Oncol. 2009 Feb;20(2):231-8. doi: 10.1093/annonc/mdn622. Epub 2008 Oct 3. PMID 18836090
- [Background] Schneider PM, Baldus SE, Metzger R, Kocher M, Bongartz R, Bollschweiler E, Schaefer H, Thiele J, Dienes HP, Mueller RP, Hoelscher AH. Histomorphologic tumor regression and lymph node metastases determine prognosis following neoadjuvant radiochemotherapy for esophageal cancer: implications for response classification. Ann Surg. 2005 Nov;242(5):684-92. doi: 10.1097/01.sla.0000186170.38348.7b. PMID 16244542
- [Result] Bollschweiler E, Holscher AH, Herbold T, Metzger R, Alakus H, Schmidt H, Drebber U, Warnecke-Eberz U. Molecular Markers for the Prediction of Minor Response to Neoadjuvant Chemoradiation in Esophageal Cancer: Results of the Prospective Cologne Esophageal Response Prediction (CERP) Study. Ann Surg. 2016 Nov;264(5):839-846. doi: 10.1097/SLA.0000000000001911. PMID 27741011